CLINICAL TRIAL: NCT06734533
Title: A New Option for Post-CDK4/6is Resistance Era: Multicenter Real-world Study of Anlotinib-based Combination Therapy in Hormone Receptor-positive Metastatic Breast Cancer Resistant to CDK4/6is.
Brief Title: Anlotinib-based Combination Therapy in Patients with Hormone Receptor-positive（HR+） Metastatic Breast Cancer(MBC) .
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ALTER-BC-005
Record Dates: First submitted 2024-11-03; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: HR+ Breast Cancer
MeSH Terms: interventions — sintilimab; Fulvestrant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Other: Anlotinib+eribulin/nab-paclitaxel/etoposide/capecitabine/pembrolizumab/ sintilimab/ fulvestrant, etc — Anlotinib (8/10/12 mg daily, Day 1-14 of each cycle) was administered orally to fasting patients, with dose reductions to 10 mg or 8 mg in cases of intolerable toxicity. Combination agents included eribulin, nab-paclitaxel, etoposide, capecitabine, pembrolizumab, sintilimab, or fulvestrant, among others.

SUMMARY:
Cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitors combined with hormonal therapy are the current standard frontline treatment for patients with hormone receptor-positive (HR+), human epidermal growth factor receptor 2 (HER-2)-negative metastatic breast cancer (MBC). However, the optimal treatment after progression on CDK4/6 inhibitors remains unknown. Anlotinib is an oral multi-target tyrosine kinase inhibitor (TKI) that strongly inhibits VEGFR, PDGFR, FGFR, and c-kit. This study aimed to evaluate the safety and efficacy of anlotinib-based combination therapy in patients with HR+ MBC previously treated with a CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 75 years, with an ECOG score of 0-1, and an expected survival of at least 3 months;
* Presence of measurable lesions as defined by RECIST 1.1 criteria;
* Histopathologically confirmed HR-positive/HER2-negative breast cancer. HER2 negativity is determined by an immunohistochemistry (IHC) result of HER2 (0/1+). If the result is HER2 (++), a FISH or CISH test is required to confirm the absence of HER2 amplification;
* Patients who have undergone multiple lines of advanced therapy with no remaining standard treatment options;
* Prior treatment with at least one line of CDK4/6 inhibitors and endocrine therapy;
* Disease progression following aromatase inhibitor (AI) or fulvestrant combined with CDK4/6 inhibitors, either as adjuvant therapy or as systemic treatment for advanced disease.

Exclusion Criteria:

* Patients with HER2-positive breast cancer confirmed by histology or cytology;
* Patients who discontinued therapy due to non-disease progression reasons, such as adverse events or other non-medical factors;
* Detection of a second primary malignant tumor at the time of enrollment;
* Failure to complete CDK4/6 inhibitor therapy;
* Pregnant or breastfeeding patients;
* Presence of third-space fluid accumulation (e.g., pleural effusion, ascites, pericardial effusion) that cannot be managed through drainage or other methods;
* Patients previously treated with anti-angiogenic agents, including small molecules such as anlotinib or apatinib, and large molecules such as bevacizumab;
* Patients currently receiving any other anti-tumor treatment for any other malignancies.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+ metastatic breast cancer previously treated with CDK4/6is
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | through study completion, an average of 1 year
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.

SECONDARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 1 year
  The ORR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)
Disease control rate (DCR) | through study completion, an average of 1 year
  The DCR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) or partial response (PR) or stable disease (SD).
Overall survival(OS) | through study completion, an average of 5 year
  OS, defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Incidence of Treatment-Emergent Adverse Events (Safety) | through study completion, an average of 1 year
  All the treatment-related adverse events occurred as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Tumor Hospital, Changsha, Hunan, China